CLINICAL TRIAL: NCT04533893
Title: Comparing Basic Life Support Performance Data Acquired From Serious Game Based Module and Simulation Based Hands on Training Via Built in Sensors of Simulators
Brief Title: Comparing Basic Life Support Performance With Serious Game Based Module and Simulation Based Hands on Training
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Emin Aksoy, Director of CASE(Center of Advamnced Simulation and Education), Acibadem University
Other Study IDs: ATADEK-2020/16
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cardiopulmonary Resuscitation; Simulation Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BLS Training Group (Students without prior BLS Training): 1. After completing training mode of the serious game module, participants were asked to choose the self-test mode of the serious game module.
  2. the participants were asked to practice their hands-on skills in simulation center under the supervision of educators. After familiarization with the system using self-training mode, the participants were asked to proceed the BLS Hands-on training app with the simulator under the supervision of the educator.
  3. Conventional OSCE score of each participant was obtained by watching the recorded sessions of BLS trainings.
  Interventions: Other: Medical simulator (3B Scientific Lilly Pro) and Platform combining simulator sensor data with OSCE scores

INTERVENTIONS:
Other: Medical simulator (3B Scientific Lilly Pro) and Platform combining simulator sensor data with OSCE scores — Hands-on training app combining OSCE scoring criteria with sensor data retrieved from the simulator's sensors was used for hands-on performance evaluation.
  Other Names: Basic Life Support Serious Game Module

SUMMARY:
The aim of this study is creating this platform and investigating whether performance evaluation of BLS trainings would be more objective compared to conventional OSCE (Objective Structured Clinical Examination) exams, if these evaluations were carried out with the platform which is combining OSCE scoring criteria with sensor data retrieved from the simulator's sensors.

DETAILED DESCRIPTION:
The participants of this study consisted of 25 volunteers among Acibadem Mehmet Ali Aydinlar University students without prior knowledge of basic life support protocol. 11 Participants (44.0%) were male, 14 (56.0%) were female. The participants were informed about the study and signed consent forms before participating the study. After a brief introduction of the serious gaming module, the participants were asked to choose the self-test mode of the serious game module. The participants' number of attempts was not limited. Following serious game based training, the hands-on training module combining OSCE scoring criteria with sensor data retrieved from the simulator's sensors was used for hands-on performance evaluation. After familiarization with the system using self-training mode, the participants were asked to proceed the BLS Hands-on training app with the simulator under the supervision of the educator. The simulation sessions were also recorded in order to use these recordings for conventional OSCE (Objective Structured Clinical Examination) performance evaluation. Conventional OSCE score of each participant was obtained by watching the recorded sessions of BLS trainings.Spearman's rho correlation test was used for calculating the correlation between serious gaming, hands on training module with including sensor data from the simulator and OSCE scores.

ELIGIBILITY:
Inclusion Criteria:

* Having no prior Basic Life Support Training

Exclusion Criteria:

* Having prior Basic Life Support Training

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants of this study consisted of 25 volunteers among Acıbadem Mehmet Ali Aydinlar University students without prior knowledge of basic life support protocol. 11 Participants (44.0%) were male, 14 (56.0%) were female. The mean age of the participants was 24,2 years.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-22 (Actual)

PRIMARY OUTCOMES:
Getting BLS(Basic Life Support Training) performance scores from serious gaming module, hands -on module with sensor data and OSCE exam on day 1. | One day
  Serious gaming module, hands -on module with sensor data and OSCE exam had the same scoring criteria depending European Resuscitation Council Basic Life Support 2015 Algorithm. The scores were calculated over 100 points, whereas higher scores meant better scores. The participants were considered as successful, if at least 80 points out of 100 were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Emin Aksoy, Ph.D., Principal Investigator — Acibadem University Case(center Of Advanced Simulation And Education)
Locations (1):
- Acibadem Mehmet Ali Aydinlar University - CASE (Center of Advanced Simulation and Education), Istanbul, Non-US/Canada, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksoy ME. Comparing Basic Life Support Serious Gaming Scores With Hands-on Training Platform Performance Scores: Pilot Simulation Study for Basic Life Support Training. JMIR Serious Games. 2020 Nov 25;8(4):e24166. doi: 10.2196/24166. PMID 33237035